CLINICAL TRIAL: NCT04414787
Title: Operationalizing PCplanner, a Needs-focused Palliative Care for Older Adults in Intensive Care Units: a Randomized Clinical Trial
Brief Title: A Needs-focused Palliative Care Intervention for Older Adults in ICUs
Acronym: PCplanner
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Pro00101745; R01AG058915 (NIH)
Record Dates: First submitted 2020-06-01; First posted 2020-06-04 (Actual); Results first posted 2025-07-18 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Palliative Care; Critical Illness; Aging; Care Delivery Model; Informal Caregivers; Psychological Distress
Keywords: palliative care; Intensive Care Unit; critical illness; mobile app; care delivery; informal caregiver
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Intervention Model Description: Randomized clinical trial comparing intervention to usual care control.
Who Masked: Participant, Outcomes Assessor
Masking Description: All masking done via differential user accesses allowed by a mobile app platform.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Active Comparator): PCplanner intervention during hospitalization
  Interventions: Behavioral: PCplanner
- Usual care control (No Intervention): Usual care

INTERVENTIONS:
Behavioral: PCplanner — PCplanner-augmented care. The PCplanner mobile app will allow patients / family members to report their needs in a platform viewable by ICU physicians. Should the needs not improve over time, the palliative care team will be activated to contribute to care.
  Arms: Intervention

SUMMARY:
The quality of intensive care unit (ICU)-based palliative care is highly variable, particularly for the 2 million older adults admitted annually to ICUs. To address these care delivery barriers among older ICU patients, a mobile app platform called PCplanner (Palliative Care planner) was developed. PCplanner automates the identification of high-risk patients (e.g., dementia, declining health status, poor functioning) by directly capturing data from electronic health record (EHR) systems, cultivates family engagement with supportive information and a digital system for self-report of actual needs, and facilitates the delivery of care to those with a high burden of need by coordinating collaboration between ICU teams and palliative care specialists.

150 patients, 150 family caregivers, and 75 physicians from academic and community settings will be enrolled in a RCT designed to test the efficacy of PCplanner-augmented collaborative palliative care vs usual care. Family caregiver and clinician experiences will be explored using mixed methods to understand intervention mechanisms as well as implementation barriers within diverse case contexts. The key hypothesis is that compared to usual care, PCplanner will reduce family caregivers' unmet needs and psychological distress, increase the frequency of goal concordant treatment among older adult patients, and reduce hospital length of stay.

DETAILED DESCRIPTION:
The quality of intensive care unit (ICU)-based palliative care is highly variable, particularly for the 2 million older adults admitted annually to ICUs. However, improving care quality on a broad scale with the efficient delivery of patient-centered, need-targeted palliative care is challenging because of logistical and technological barriers. To address these care delivery barriers among older ICU patients, a mobile app platform called PCplanner (Palliative Care planner) was developed. PCplanner automates the identification of high-risk patients (e.g., dementia, declining health status, poor functioning) by directly capturing data from electronic health record (EHR) systems, cultivates family engagement with supportive information and a digital system for self-report of actual needs, and facilitates the delivery of care to those with a high burden of need by coordinating collaboration between ICU teams and palliative care specialists. In pilot comparison to a standard palliative care control, the intervention reduced unmet needs, psychological distress, and length of stay and increased goal concordant care, communication, and hospice utilization.

While these data are compelling, an efficacy evaluation of PCplanner is needed. Therefore, we plan to enroll approximately 150 patients, 150 family caregivers, and 75 physicians will be enrolled from academic and community settings in a project with 2 key aims: (1) Test the efficacy of PCplanner-augmented collaborative palliative care vs usual care in a randomized clinical trial (RCT) with 3-month follow up, and (2) Explore family caregiver and clinician experiences using mixed methods to understand intervention mechanisms as well as implementation barriers within diverse case contexts. The key hypothesis is that compared to usual care, PCplanner will reduce family caregivers' unmet needs and psychological distress, increase the frequency of goal concordant treatment among older adult patients, and reduce hospital length of stay.

ELIGIBILITY:
PATIENTS

Inclusion Criteria:

* ≥50 years of age
* Receive care in a study ICU for ≥24 hours
* Meets ≥1 of 9 high risk phenotypes a. Dementia (e.g., Alzheimer's, multi-infarct, other dementia etiology) b. Declining health status defined by EITHER: i. ≥2 hospital admissions in 3 months preceding current admission OR ii. >1 ICU admission in 3 months preceding current admission c. Poor functional status defined by EITHER: i. admit from Skilled Nursing Facility (SNF) or Long-Term Acute Care (LTAC) facility OR ii. ≥3 activities of daily living (ADL) limitations at admission d. Severe acute illness defined by EITHER: i. cardiac arrest OR ii. multisystem organ failure (≥3 of: lung, kidney, hematological, brain, cardiac, liver) that has worsened over 48 hours (i.e., Sequential Organ Failure Assessment [SOFA] score increase) e. Severe acute stroke (e.g., acute intracranial hemorrhage, ischemic stroke, or traumatic brain injury) f. Acute respiratory failure (ventilation or high oxygen support for ≥24 hours) g. Acute renal failure (new hemodialysis or continuous venovenous hemodiafiltration for ≥1 hour) h. Advanced cancer (Advanced / metastatic cancer diagnosis) i. Shock (use of vasopressor or inotrope for ≥4 hours)

Exclusion Criteria (pre-consent):

* Palliative care consultation performed during the hospitalization before eligibility determination
* Current admission to ICU at the index hospital ≥8 days
* Imprisoned
* No known family or surrogate decision maker
* Death expected within 24 hours

Exclusion Criteria (post-consent):

- Patient dies before T2

FAMILY MEMBER

Inclusion Criteria:

* ≥18 years of age
* Self-described as the individual (related or unrelated) who provides the most support and with whom the patient has a significant relationship (per definition of 'family' described in the Society of Critical Care Medicine 2016 Guidelines for Family-Centered Care in the Neonatal, Pediatric, and Adult ICU)

Exclusion Criteria (pre-consent):

* Lack a knowledge of English such that the potential participant is not confident that they could complete study tasks (app viewing, surveys)
* Imprisoned
* Unable to complete surveys for any reason

Exclusion Criteria (post-consent):

- Low need burden (NEST score <10) at baseline

ICU PHYSICIANS

Inclusion Criteria:

* ≥18 years of age
* Attending or fellow physician in a study ICU

Exclusion Criteria:

- None

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2021-02-22 (Actual); Primary Completion 2023-09-26 (Actual); Study Completion 2023-12-17 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Cox, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Per NIH and Duke University policies after trial and analyses completed.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 2025
Access Criteria: review by study team

REFERENCES:
- [Background] Cox CE, Jones DM, Reagan W, Key MD, Chow V, McFarlin J, Casarett D, Creutzfeldt CJ, Docherty SL. Palliative Care Planner: A Pilot Study to Evaluate Acceptability and Usability of an Electronic Health Records System-integrated, Needs-targeted App Platform. Ann Am Thorac Soc. 2018 Jan;15(1):59-68. doi: 10.1513/AnnalsATS.201706-500OC. PMID 29121480
- [Background] Cox CE, Olsen MK, Casarett D, Haines K, Al-Hegelan M, Bartz RR, Katz JN, Naglee C, Ashana D, Gilstrap D, Gu J, Parish A, Frear A, Krishnamaneni D, Corcoran A, Docherty SL. Operationalizing needs-focused palliative care for older adults in intensive care units: Design of and rationale for the PCplanner randomized clinical trial. Contemp Clin Trials. 2020 Nov;98:106163. doi: 10.1016/j.cct.2020.106163. Epub 2020 Sep 29. PMID 33007442
- [Derived] Cox CE, Ashana DC, Dempsey K, Olsen MK, Parish A, Casarett D, Johnson KS, Haines KL, Naglee C, Katz JN, Al-Hegelan M, Riley IL, Docherty SL. Mobile App-Facilitated Collaborative Palliative Care Intervention for Critically Ill Older Adults: A Randomized Clinical Trial. JAMA Intern Med. 2025 Feb 1;185(2):173-183. doi: 10.1001/jamainternmed.2024.6838. PMID 39680398
- See also: general trial information — http://pcplanner.duke.edu

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1. Physicians and patients were not considered enrolled for study measure purposes as NEITHER completed surveys or other self-reported outcomes. 2. Physicians were not randomized to a group and therefore cannot be sensibly included in a RCT data table. 3. Note in the flow table these are also the numbers of patient-family members dyads. ONLY FAMILY MEMBERS completed surveys in this trial. They are not represented in separate flow diagrams because it would be too confusing for the reader.
Groups:
- PCplanner Intervention Dyad - Family Member; PCplanner Intervention Dyad - Patient: PCplanner intervention during hospitalization
  PCplanner: PCplanner-augmented care. The PCplanner mobile app will allow patients' family members to report their needs in a platform viewable by ICU physicians. Should the needs not improve over time, the palliative care team will be activated to contribute to care.
- Usual Care Control Dyad - Family Member; Usual Care Control Dyad - Patient: Usual care includes standard ICU care
Period: Overall Study
Arm/Group | PCplanner Intervention Dyad - Family Member | PCplanner Intervention Dyad - Patient | Usual Care Control Dyad - Family Member | Usual Care Control Dyad - Patient
Started | 76 | 76 | 75 | 75
Completed (Deaths and hospitalizations reflect patients, not family members/caregivers. Those patients' caregivers were not able to complete the study.) | 47 | 47 | 48 | 48
Not Completed | 29 | 29 | 27 | 27
Not completed — Patient Death | 18 | 18 | 15 | 15
Not completed — Patient Hospitalization | 1 | 1 | 2 | 2
Not completed — Lost to Follow-up | 7 | 7 | 5 | 5
Not completed — Residence in post-acute care facility | 3 | 3 | 5 | 5

BASELINE CHARACTERISTICS:
Population: ONLY FAMILY MEMBERS have survey outcomes reported (i.e., NEST). Physicians and patients DID NOT complete surveys.
  The ONLY patient-level data reported are for demographics, length of stay, and AEs.
Groups:
- PCplanner Intervention Family Members; PCplanner Intervention Patients: PCplanner intervention during hospitalization
  PCplanner: PCplanner-augmented care. The PCplanner mobile app will allow patients' family members to report their needs in a platform viewable by ICU physicians. Should the needs not improve over time, the palliative care team will be activated to contribute to care.
- Usual Care Control Family Members; Usual Care Control Patients: Usual care is standard ICU care
- Total: Total of all reporting groups
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members | PCplanner Intervention Patients | Usual Care Control Patients | Total
Number analyzed (Participants) | 76 | 75 | 76 | 75 | 302
Age, Continuous [Mean (Standard Deviation); unit: years] | 57.3 (12.9) | 57.4 (13.0) | 69.2 (9.8) | 70.5 (9.6) | 57.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 53 | 57 | 34 | 31 | 175
  Male | 23 | 18 | 42 | 44 | 127
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 1 | 1 | 4
  Not Hispanic or Latino | 74 | 74 | 75 | 73 | 296
  Unknown or Not Reported | 1 | 0 | 0 | 1 | 2
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 2 | 0 | 2 | 4
  Native Hawaiian or Other Pacific Islander | 0 | 1 | 0 | 0 | 1
  Black or African American | 23 | 14 | 23 | 14 | 74
  White | 50 | 56 | 52 | 58 | 216
  More than one race | 0 | 1 | 0 | 1 | 2
  Unknown or Not Reported | 3 | 0 | 1 | 0 | 4
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 76 | 75 | 76 | 75 | 302
NEST score [Mean (Standard Deviation); unit: units on a scale] — The NEST (Needs; Existential Concerns; Symptoms; and Therapeutic Interaction) is a palliative care needs instrument capturing all 8 domains of palliative care quality. Scores range from 0 (no needs) to 130 (higher needs).
  Note that NEST data were not captured from patients. On family members completed the NEST. Population: NEST surveys were not collected from patients.
  units on a scale
    number analyzed (Participants) | 76 | 75 | 0 | 0 | 151
    (all) | 31.8 (18.4) | 32.6 (17.9) |  |  | 32.2 (18.1)

OUTCOME MEASURES:

1. Primary Outcome: Needs; Existential Concerns; Symptoms; and Therapeutic Interaction (NEST) Scale Total Score
Description: The NEST is a palliative care needs instrument capturing all 8 domains of palliative care quality from patients' family members. Scores range from 0 (no needs) to 130 (higher needs). Reported here is scores at Time 3 (~1 week post-randomization).
Time Frame: Time 1 (baseline), Time 2 (~3 days post-randomization), and Time 3 (~1 week post-randomization)
Population: Participants with data collected at Time 3 (~1 week post-randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 61 | 53
score on a scale | 28.5 (19.4) | 29.3 (21.4)
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Difference between Time 1 (baseline) and Time 3 (~1 week post-randomization); Test type: Superiority; p = 1.00, Mixed Models Analysis; Mean Difference (Final Values) = 0.0, 95% CI 2-sided [-6.21 to 6.21]

2. Secondary Outcome: Patient Health Questionnaire 9-Item Scale (PHQ-9)
Description: A depression symptoms instrument used by patients' family members. Scores range from 0 (no depression symptoms) to 27 (higher depression symptoms). Reported here is the scores at Time 4 (3 months post-randomization).
Time Frame: Time 1 (baseline), Time 3 (~1 week post-randomization), and Time 4 (3 months post-randomization)
Population: Participants with data collected at Time 4 (3 months post-randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 47 | 48
score on a scale | 6.0 (4.6) | 6.3 (5.3)
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Difference between Time 1 (baseline) and Time 4 (3 months post-randomization); Test type: Superiority; p = 0.95, Mixed Models Analysis; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-1.83 to 1.72]

3. Secondary Outcome: Generalized Anxiety Disorder 7-Item Scale (GAD-7)
Description: An anxiety symptoms instrument used by patients' family members. Scores range from 0 (no anxiety symptoms) to 21 (higher anxiety symptoms). Reported here is the scores at Time 4 (3 months post-randomization).
Time Frame: Time 1 (baseline), Time 3 (target ~1 week post-randomization), and Time 4 (3 months post-randomization)
Population: Participants with data collected at Time 4 (3 months post-randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 47 | 48
score on a scale | 4.9 (5.2) | 4.8 (3.9)
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Difference between Time 1 (baseline) and Time 4 (3 months post-randomization); Test type: Superiority; p = 0.72, Mixed Models Analysis; Mean Difference (Final Values) = 0.29, 95% CI 2-sided [-1.28 to 1.86]

4. Secondary Outcome: Post-Traumatic Stress Symptom (PTSS) Inventory
Description: A post-traumatic stress disorder symptom instrument used by patients' family members. Scores range from 10 (low PTSD symptoms) to 70 (higher PTSD symptoms). Reported here is the scores at Time 4 (3 months post-randomization).
Time Frame: Time 1 (baseline) and Time 4 (3 months post-randomization)
Population: Participants with data collected at Time 4 (3 months post-randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 47 | 48
score on a scale | 21.7 (13.1) | 21.6 (11.3)
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Difference between Time 1 (baseline) and Time 4 (3 months post-randomization); Test type: Superiority; p = 0.48, Mixed Models Analysis; Mean Difference (Final Values) = 1.35, 95% CI 2-sided [-2.44 to 5.14]

5. Secondary Outcome: Number of Participants With Goal Concordant Care
Description: A metric of goal concordance as reported by patients' family members.
Time Frame: Time 1 (baseline), Time 2 (target ~3 days post-randomization), and Time 3 (target ~1 week post-randomization)
Population: Participants with data collected at Time 3 (~1 week post-randomization).
Measure: Count of Participants; unit: Participants
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 61 | 53
Participants | 49 | 45
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Difference between Time 1 (baseline) and Time 3 (target ~1 week post-randomization); Test type: Superiority; p = 0.12, Mixed Models Analysis; Odds Ratio (OR) = 0.49, 95% CI 2-sided [0.20 to 1.2]

6. Secondary Outcome: Patient-Perceived Patient-Centeredness (PPPC) Scale
Description: A measure of patient-centeredness used by patients' family members with scores that range from 12 (higher patient-centeredness) to 48 (lower patient-centeredness).
Time Frame: Time 3 (target ~1 week post-randomization)
Population: Participants with data collected at Time 3 (~1 week post-randomization).
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members
Number analyzed (Participants) | 61 | 53
score on a scale | 20.2 (7.0) | 21.4 (8.4)
Statistical Analysis 1: Comparison: PCplanner Intervention Family Members vs Usual Care Control Family Members; Test type: Superiority; p = 0.58, Wilcoxon (Mann-Whitney)

7. Secondary Outcome: Post-randomization Intensive Care Unit Length of Stay
Description: A measure of intensive care unit days after randomization for patients of whom participants are family members/caregivers.
Time Frame: from randomization until intensive care unit discharge
Population: Patients of whom participants are family members/caregivers.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PCplanner Intervention Patients | Usual Care Control Patients
Number analyzed (Participants) | 76 | 75
days | 11.5 [6.0 to 60.0] | 10.0 [7.0 to 23.0]
Statistical Analysis 1: Comparison: PCplanner Intervention Patients vs Usual Care Control Patients; Test type: Superiority; p = 0.29, Wilcoxon (Mann-Whitney)

8. Secondary Outcome: Post-randomization Hospital Length of Stay
Description: A measure of hospital days after randomization for PATIENTS for each patient member of the patient-family member dyad
Time Frame: from randomization until hospital discharge
Population: Patients of whom participants are family members/caregivers.
Measure: Median (Inter-Quartile Range); unit: days
Arm/Group | PCplanner Intervention Patients | Usual Care Control Patients
Number analyzed (Participants) | 76 | 75
days | 19.0 [12.0 to 31.0] | 20.0 [12.0 to 32.0]
Statistical Analysis 1: Comparison: PCplanner Intervention Patients vs Usual Care Control Patients; Test type: Superiority; p = 0.79, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 3 months
Description: Adverse event reporting by family members and patients are as follows. Numbers reported for PHQ-9 item 9 (suicidality) reflect FAMILY MEMBERS. Numbers reported for deaths reflect PATIENTS.
Groups:
- PCplanner Intervention Family Members: PCplanner intervention during hospitalization
  PCplanner: PCplanner-augmented care. The PCplanner mobile app will allow patients / family members to report their needs in a platform viewable by ICU physicians. Should the needs not improve over time, the palliative care team will be activated to contribute to care.
  Adverse event reporting by family members and patients are as follows. Numbers reported for PHQ-9 item 9 (suicidality) reflect FAMILY MEMBERS.
- Usual Care Control Family Members: Usual care is standard ICU care
  Adverse event reporting by family members and patients are as follows. Numbers reported for PHQ-9 item 9 (suicidality) reflect FAMILY MEMBERS.
- PCplanner Intervention Patients: PCplanner intervention during hospitalization
  PCplanner: PCplanner-augmented care. The PCplanner mobile app will allow patients / family members to report their needs in a platform viewable by ICU physicians. Should the needs not improve over time, the palliative care team will be activated to contribute to care.
  Adverse event reporting by family members and patients are as follows. Numbers reported for deaths reflect PATIENTS.
- Usual Care Control Patients: Usual care is standard ICU care
  Adverse event reporting by family members and patients are as follows. Numbers reported for deaths reflect PATIENTS.
Arm/Group | PCplanner Intervention Family Members | Usual Care Control Family Members | PCplanner Intervention Patients | Usual Care Control Patients
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/75 | 18/76 | 15/75
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/75 | 0/76 | 0/75
Other Adverse Events (participants affected / at risk) | 1/76 | 1/75 | 0/76 | 0/75
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PCplanner Intervention Family Members (N=76) | Usual Care Control Family Members (N=75) | PCplanner Intervention Patients (N=76) | Usual Care Control Patients (N=75)
Family member reporting a value other than 1 for PHQ-9 item 9 (suicidality) (Psychiatric disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0) — Note PI called both participant immediately to ensure safety and confirm there was no active suicidality.

LIMITATIONS AND CAVEATS:
Deaths reported reflect patient, not family member, events.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2022-06-13): https://cdn.clinicaltrials.gov/large-docs/87/NCT04414787/Prot_SAP_001.pdf
  • Informed Consent Form (2022-12-05): https://cdn.clinicaltrials.gov/large-docs/87/NCT04414787/ICF_000.pdf